CLINICAL TRIAL: NCT01732757
Title: A Study to Evaluate the Efficacy of Lastacaft® Compared to Pataday™ and Placebo in Patients With Acute Allergic Conjunctivitis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GMA-LAS-12-023
Record Dates: First submitted 2012-11-19; First posted 2012-11-26 (Estimated); Results first posted 2014-01-14 (Estimated); Last update posted 2014-01-14 (Estimated); Status verified 2013-11

CONDITIONS: Conjunctivitis, Allergic
MeSH Terms: conditions — Conjunctivitis, Allergic | interventions — alcaftadine; Olopatadine Hydrochloride; Dextrans; Lubricant Eye Drops

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Lastacaft® (Active Comparator): One drop of Lastacaft® (Alcaftadine 0.25%) administered in both eyes on Day 0.
  Interventions: Drug: Alcaftadine 0.25%
- Pataday™ (Active Comparator): One drop of Pataday™ (Olopatadine 0.2%) administered in both eyes on Day 0.
  Interventions: Drug: Olopatadine 0.2%
- Placebo (dextran 70 0.1%/hydroxypropyl methylcellulose 0.3%) (Placebo Comparator): One drop of Placebo (dextran 70 0.1%/hydroxypropyl methylcellulose 0.3%) administered in both eyes on Day 0.
  Interventions: Drug: dextran 70 0.1%/hydroxypropyl methylcellulose 0.3%

INTERVENTIONS:
Drug: Alcaftadine 0.25% — One drop of Lastacaft® (Alcaftadine 0.25%) administered in both eyes on Day 0.
  Other Names: Lastacaft®
  Arms: Lastacaft®
Drug: Olopatadine 0.2% — One drop of Pataday™ (Olopatadine 0.2%) administered in both eyes on Day 0.
  Other Names: Pataday™
  Arms: Pataday™
Drug: dextran 70 0.1%/hydroxypropyl methylcellulose 0.3% — One drop of placebo (dextran 70 0.1%/hydroxypropyl methylcellulose 0.3%) administered in both eyes on Day 0.
  Other Names: Tears Naturale II
  Arms: Placebo (dextran 70 0.1%/hydroxypropyl methylcellulose 0.3%)

SUMMARY:
This study will evaluate the efficacy of Lastacaft® (Alcaftadine 0.25%) and Pataday™ (Olopatadine 0.2%) as compared to each other and to placebo in the prevention of ocular itching associated with allergic conjunctivitis.

ELIGIBILITY:
Inclusion Criteria:

* History of ocular allergies within the past 24 months.
* Able to avoid wearing contact lenses for at least 72 hours prior to and during the study trial period.

Exclusion Criteria:

* Any presence of active ocular infection or history of an ocular herpetic infection.
* Ocular surgery within 3 months prior to the first visit or refractive surgery within the past 6 months.
* Have any planned surgery during the study or 30 days after the study.

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 157 (Actual)
Dates: Start 2012-11; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan
Locations (1):
- Memphis, Tennessee, United States

REFERENCES:
- [Derived] McLaurin EB, Marsico NP, Ackerman SL, Ciolino JB, Williams JM, Villanueva L, Hollander DA. Ocular itch relief with alcaftadine 0.25% versus olopatadine 0.2% in allergic conjunctivitis: pooled analysis of two multicenter randomized clinical trials. Adv Ther. 2014 Oct;31(10):1059-71. doi: 10.1007/s12325-014-0155-3. Epub 2014 Sep 27. PMID 25260889

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Lastacaft® | Pataday™ | Placebo (Dextran 70 0.1%/Hydroxypropyl Methylcellulose 0.3%)
Started | 53 | 52 | 52
Completed | 52 | 52 | 52
Not Completed | 1 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lastacaft® | Pataday™ | Placebo (Dextran 70 0.1%/Hydroxypropyl Methylcellulose 0.3%) | Total
Number analyzed (Participants) | 53 | 52 | 52 | 157
Age, Continuous [Mean (Standard Deviation); unit: Years] | 38.2 (13.78) | 38.7 (15.10) | 34.7 (12.58) | 37.2 (13.88)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 29 | 26 | 87
  Male | 21 | 23 | 26 | 70

OUTCOME MEASURES:

1. Primary Outcome: Ocular Itching Evaluated by the Subject 3 Minutes Post Challenge on Day 0
Description: Ocular itching is evaluated by the subject at 3 minutes post challenge on Day 0 (Visit 3B). Subjects score their ocular itching on a 9-point numeric analog scale ranging from 0=None to 4=Incapacitating Itch with an Irresistible Urge to Rub (0.5 increments are allowed). For each subject, the score for both eyes is averaged (i.e., one score per subject). A lower score is indicative of less itching.
Time Frame: Day 0 at 3 Minutes Post Challenge
Population: All randomized subjects with data at this time point
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | Lastacaft® | Pataday™ | Placebo (Dextran 70 0.1%/Hydroxypropyl Methylcellulose 0.3%)
Number analyzed (Participants) | 52 | 52 | 52
Scores on a Scale | 0.40 (0.582) | 0.76 (0.752) | 2.00 (1.109)

2. Secondary Outcome: Ocular Itching Evaluated by the Subject at 5 and 7 Minutes Post Challenge on Day 0
Description: Ocular itching is evaluated by the subject at 5 and 7 minutes post challenge on Day 0 (Visit 3B). Subjects score their ocular itching on a 9-point numeric analog scale ranging from 0=None to 4=Incapacitating Itch with an Irresistible Urge to Rub (0.5 increments are allowed). For each subject, the score for both eyes is averaged (i.e., one score per subject). A lower score is indicative of less itching.
Time Frame: Day 0
Population: All randomized subjects with data at this time point
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | Lastacaft® | Pataday™ | Placebo (Dextran 70 0.1%/Hydroxypropyl Methylcellulose 0.3%)
Number analyzed (Participants) | 52 | 52 | 52
Scores on a Scale
  5 Minutes | 0.61 (0.663) | 0.79 (0.725) | 2.08 (1.061)
  7 Minutes | 0.69 (0.724) | 0.71 (0.774) | 1.89 (1.114)

3. Secondary Outcome: Percentage of Subjects With Minimal Itching Score at 3, 5, and 7 Minutes Post Challenge on Day 0
Description: Ocular itching is evaluated by the subject at 3, 5, and 7 minutes post challenge on Day 0 (Visit 3B). Subjects score their ocular itching on a 9-point numeric analog scale ranging from 0=None to 4=Incapacitating Itch with an Irresistible Urge to Rub (0.5 increments are allowed). For each subject, the score for both eyes is averaged (i.e., one score per subject). Minimal itching is considered a score <1.
Time Frame: Day 0
Population: All randomized subjects with data at this time point
Measure: Number; unit: Percentage of Subjects
Arm/Group | Lastacaft® | Pataday™ | Placebo (Dextran 70 0.1%/Hydroxypropyl Methylcellulose 0.3%)
Number analyzed (Participants) | 52 | 52 | 52
Percentage of Subjects
  3 Minutes | 84.6 | 65.4 | 21.2
  5 Minutes | 75.0 | 53.8 | 21.2
  7 Minutes | 69.2 | 61.5 | 25.0

4. Secondary Outcome: Percentage of Subjects With a Zero Itch Score at 3, 5, and 7 Minutes Post Challenge on Day 0
Description: Ocular itching is evaluated by the subject at 3, 5, and 7 minutes post challenge on Day 0 (Visit 3B). Subjects score their ocular itching on a 9-point numeric analog scale ranging from 0=None to 4=Incapacitating Itch with an Irresistible Urge to Rub (0.5 increments are allowed). For each subject, the score for both eyes is averaged (i.e., one score per subject). Zero itch is considered a score = 0.
Time Frame: Day 0
Population: All randomized subjects with data at this time point
Measure: Number; unit: Percentage of Subjects
Arm/Group | Lastacaft® | Pataday™ | Placebo (Dextran 70 0.1%/Hydroxypropyl Methylcellulose 0.3%)
Number analyzed (Participants) | 52 | 52 | 52
Percentage of Subjects
  3 Minutes | 48.1 | 26.9 | 5.8
  5 Minutes | 26.9 | 26.9 | 3.8
  7 Minutes | 26.9 | 32.7 | 7.7

5. Secondary Outcome: Percentage of Subject Eyes in Each Category of the Itching Score Distribution Post Challenge on Day 0
Description: Ocular itching is evaluated by the subject at Hour 16 post challenge on Day 0. Subjects score their ocular itching on a 9-point numeric analog scale ranging from 0=None to 4=Incapacitating Itch with an Irresistible Urge to Rub (0.5 increments are allowed).
Time Frame: Day 0
Population: All randomized subjects with data at this time point
Measure: Number; unit: Percentage of Subject Eyes
Units Other Than Participants: Eyes
Arm/Group | Lastacaft® | Pataday™ | Placebo (Dextran 70 0.1%/Hydroxypropyl Methylcellulose 0.3%)
Number analyzed (Participants) | 52 | 52 | 52
Number analyzed (Eyes) | 104 | 104 | 104
Percentage of Subject Eyes
  0 | 41.7 | 34.3 | 8.7
  0.5 | 32.1 | 24.0 | 10.9
  1.0 | 12.5 | 20.8 | 8.0
  1.5 | 3.5 | 7.7 | 6.4
  2.0 | 5.8 | 6.7 | 17.9
  2.5 | 4.2 | 5.1 | 22.8
  3.0 | 0.3 | 1.3 | 15.1
  3.5 | 0.0 | 0.0 | 5.8
  4.0 | 0.0 | 0.0 | 4.5

6. Secondary Outcome: Conjunctival Redness Evaluated by the Investigator at 7, 15, and 20 Minutes Post Challenge on Day 0
Description: The conjunctiva is a thin membrane that covers the inner surface of the eyelid and the white part of the eye. Conjunctival redness is evaluated by the investigator at 7, 15, and 20 minutes post challenge on Day 0 (Visit 3B). Investigators score conjunctival redness on a 9-point numeric analog scale ranging from 0=None to 4=Extremely Severe (0.5 increments are allowed). For each subject, the score for both eyes is averaged (i.e., one score per subject). A lower score is indicative of less conjunctival redness.
Time Frame: Day 0
Population: All randomized subjects with data at this time point
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | Lastacaft® | Pataday™ | Placebo (Dextran 70 0.1%/Hydroxypropyl Methylcellulose 0.3%)
Number analyzed (Participants) | 52 | 52 | 52
Scores on a Scale
  7 Minutes | 1.73 (0.887) | 1.61 (0.867) | 2.17 (0.731)
  15 Minutes | 2.02 (0.844) | 1.81 (0.877) | 2.17 (0.784)
  20 Minutes | 2.10 (0.854) | 1.89 (0.886) | 2.22 (0.830)

7. Secondary Outcome: Ciliary Redness Evaluated by the Investigator at 7, 15, and 20 Minutes Post Challenge on Day 0
Description: Ciliary redness is redness spreading out around the cornea of the eye. Ciliary redness is evaluated by the investigator at 7, 15, and 20 minutes post challenge on Day 0 (Visit 3B). Investigators score ciliary redness on a 9-point numeric analog scale ranging from 0=None to 4=Extremely Severe (0.5 increments are allowed). For each subject, the score for both eyes is averaged (i.e., one score per subject). A lower score is indicative of less ciliary redness.
Time Frame: Day 0
Population: All randomized subjects with data at this time point
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | Lastacaft® | Pataday™ | Placebo (Dextran 70 0.1%/Hydroxypropyl Methylcellulose 0.3%)
Number analyzed (Participants) | 52 | 52 | 52
Scores on a Scale
  7 Minutes | 1.62 (0.889) | 1.47 (0.887) | 2.10 (0.805)
  15 Minutes | 1.97 (0.845) | 1.71 (0.912) | 2.12 (0.832)
  20 Minutes | 2.06 (0.831) | 1.78 (0.913) | 2.13 (0.903)

8. Secondary Outcome: Episcleral Redness Evaluated by the Investigator at 7, 15, and 20 Minutes Post Challenge on Day 0
Description: The episclera is the tissue that lies over the white part of the eye. Episcleral redness is evaluated by the investigator at 7, 15, and 20 minutes post challenge on Day 0 (Visit 3B). Investigators score episcleral redness on a 9-point numeric analog scale ranging from 0=None to 4=Extremely Severe (0.5 increments are allowed). For each subject, the score for both eyes is averaged (i.e., one score per subject). A lower score is indicative of less episcleral redness.
Time Frame: Day 0
Population: All randomized subjects with data at this time point
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | Lastacaft® | Pataday™ | Placebo (Dextran 70 0.1%/Hydroxypropyl Methylcellulose 0.3%)
Number analyzed (Participants) | 52 | 52 | 52
Scores on a Scale
  7 Minutes | 1.61 (0.842) | 1.53 (0.815) | 2.04 (0.755)
  15 Minutes | 1.88 (0.820) | 1.70 (0.839) | 2.04 (0.828)
  20 Minutes | 1.97 (0.837) | 1.78 (0.874) | 2.09 (0.837)

9. Secondary Outcome: Chemosis Evaluated by the Investigator at 7, 15, and 20 Minutes Post Challenge on Day 0
Description: Chemosis is swelling of the tissue that lines the eyelids and surface of the eye. Chemosis is evaluated by the investigator at 7, 15, and 20 minutes post challenge on Day 0 (Visit 3B). Investigators score chemosis on a 9-point numeric analog scale ranging from 0=None to 4=Severe (0.5 increments are allowed). For each subject, the score for both eyes is averaged (i.e., one score per subject). A lower score is indicative of less chemosis.
Time Frame: Day 0
Population: All randomized subjects with data at this time point
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | Lastacaft® | Pataday™ | Placebo (Dextran 70 0.1%/Hydroxypropyl Methylcellulose 0.3%)
Number analyzed (Participants) | 52 | 52 | 52
Scores on a Scale
  7 Minutes | 0.37 (0.433) | 0.27 (0.350) | 0.51 (0.511)
  15 Minutes | 0.62 (0.576) | 0.51 (0.562) | 0.76 (0.691)
  20 Minutes | 0.73 (0.679) | 0.56 (0.634) | 0.96 (0.757)

10. Secondary Outcome: Eyelid Swelling Evaluated by the Subject at 7, 15, and 20 Minutes Post Challenge on Day 0
Description: Eyelid swelling is evaluated by the subject at 7, 15, and 20 minutes post challenge on Day 0 (Visit 3B). Subjects score eyelid swelling on a 4-point numeric analog scale ranging from 0=None to 3=Severe. For each subject, the score for both eyes is averaged (i.e., one score per subject). A lower score is indicative of less lid swelling.
Time Frame: Day 0
Population: All randomized subjects with data at this time point
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | Lastacaft® | Pataday™ | Placebo (Dextran 70 0.1%/Hydroxypropyl Methylcellulose 0.3%)
Number analyzed (Participants) | 52 | 52 | 52
Scores on a Scale
  7 Minutes | 0.2 (0.48) | 0.3 (0.54) | 0.8 (0.70)
  15 Minutes | 0.4 (0.51) | 0.5 (0.70) | 0.9 (0.78)
  20 Minutes | 0.4 (0.51) | 0.6 (0.85) | 0.7 (0.76)

11. Secondary Outcome: Tearing Evaluated by the Subject at 7, 15, and 20 Minutes Post Challenge on Day 0
Description: Tearing is evaluated by the subject at 7, 15, and 20 minutes post challenge on Day 0 (Visit 3B). Subjects score tearing on a 5-point numeric analog scale ranging from 0=None/Normal to 4=Very Severe. For each subject, the score for both eyes is averaged (i.e., one score per subject). A lower score is indicative of less tearing.
Time Frame: Day 0
Population: All randomized subjects with data at this time point
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | Lastacaft® | Pataday™ | Placebo (Dextran 70 0.1%/Hydroxypropyl Methylcellulose 0.3%)
Number analyzed (Participants) | 52 | 52 | 52
Scores on a Scale
  7 Minutes | 0.2 (0.40) | 0.4 (0.59) | 0.9 (0.84)
  15 Minutes | 0.4 (0.58) | 0.5 (0.77) | 0.8 (0.93)
  20 Minutes | 0.3 (0.57) | 0.6 (0.83) | 0.7 (0.94)

ADVERSE EVENTS:
Arm/Group | Lastacaft® | Pataday™ | Placebo (Dextran 70 0.1%/Hydroxypropyl Methylcellulose 0.3%)
Serious Adverse Events (participants affected / at risk) | 0/53 | 0/52 | 0/52
Other Adverse Events (participants affected / at risk) | 0/53 | 0/52 | 0/52

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.